CLINICAL TRIAL: NCT02764372
Title: Serious Games for Upper Extremity Rehabilitation for Patients With Neurological Disorders: A Pilot Study
Brief Title: Telerehabilitation Upper Extremity for Neurological Disorders
Acronym: Telerehab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Bremen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rehab2016
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis; Stroke
Keywords: Arm rehabilitation; Serious games; stroke; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Stroke | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Serious games (Experimental): The experimental group received Serious Games-based upper extremity therapy through Kinect
  Interventions: Behavioral: Serious games
- Exergames (Active Comparator): The control played the same amount of time with commercial exergames of the Wii
  Interventions: Behavioral: Exergames

INTERVENTIONS:
Behavioral: Serious games — Participants played serious games developed for Kinect in the the EU FP7 STREP Project REHAB@HOME N. 306113
  Other Names: virtual reality games
  Arms: Serious games
Behavioral: Exergames — Participants played exergames existent in the Wii game console
  Other Names: Wii game console
  Arms: Exergames

SUMMARY:
The aims of the present study were to:

* Investigate the feasibility of using a therapeutic gaming system (REHAB@HOME), based on Kinect, to augment upper extremity neurorehabilitation services.
* Provide preliminary evidence of clinical efficacy of the approach in increasing arm activity and health related quality of life of persons post stroke or with MS.

Main results suggest that the serious games approach was positively received in terms of user experience and motivation to use, with the participants showing also improvements in functional abilities of the treated arm.

DETAILED DESCRIPTION:
The objective of this pilot study was to assess the feasibility of using a therapeutic gaming system (REHAB@HOME), based on Kinect, to augment upper extremity neurorehabilitation services. A secondary objective was to provide preliminary evidence of clinical efficacy of the approach in increasing arm activity and health related quality of life of persons post stroke or with multiple sclerosis (MS).

A pilot single-blind randomized controlled trial was carried out in an inpatient and ambulatory care at a rehabilitation center. Twenty persons with multiple sclerosis (n=16) or chronic poststroke (n=4) receiving rehabilitation at the center, able to flex shoulder and elbow at least 45 degrees, participated in the study.

An intervention group received Serious Games-based upper extremity therapy for a total of 12 sessions (4-5 sessions, lasting 40 minutes, per week) and the control played the same amount of time with commercial exergames of the Wii. Both groups received their usual rehabilitation services as well as game playing.

ELIGIBILITY:
Inclusion Criteria:

* Persons Post stroke or with MS with resultant upper extremity motor deficits.
* Range of motion of shoulder and elbow equal or higher than 45 degrees.
* Able to comprehend and follow directions.

Exclusion Criteria:

* Wearing pace maker
* Comorbidities affecting arm use
* Not able to comprehend and follow directions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
9 Hole peg test | 10 months
  Testing pre and post intervention
Box and Block test | 10 months
  Testing pre and post intervention

SECONDARY OUTCOMES:
Short Form 12 | 10 months
  Testing pre and post intervention
the EQ-5D visual analogue scale (EQ-VAS) | 10 months
  Testing pre and post intervention

IPD SHARING:
Plan to Share IPD: Undecided